CLINICAL TRIAL: NCT00838071
Title: Evaluation of Anti-Hepatitis B Antibodies Levels in Serum After the Intravenous Administration of Specific Anti-Hepatitis B Immunoglobulin (IGIV-HB Grifols) in Patients Having Previously Undergone Liver Transplantation
Brief Title: Evaluation of Serum Levels and Pharmacokinetics of a New Hepatitis B Immune Globulin Following Liver Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Antonio Páez, MD, Instituto Grifols
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IG301
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B; HBV; Anti-hepatitis B antibodies; Immunoglobulins; liver transplantation; Protective levels; Recurrence; Intravenous
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IGIV-HB Grifols (Experimental)
  Interventions: Drug: Specific intravenous anti-hepatitis B immunoglobulin

INTERVENTIONS:
Drug: Specific intravenous anti-hepatitis B immunoglobulin — Monthly doses of 5000 IU administered intravenously during 6 consecutive months
  Other Names: Niuliva

SUMMARY:
The purpose of this study is to determine whether protective anti-HB serum levels are maintained after 6 months of uninterrupted treatment with IGIV-HB Grifols, a new specific hepatitis B immune globulin, in patients having previously undergone liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having undergone a liver transplantation due to liver disease associated with hepatitis B virus, at least 1 year before and no more than 5 years before inclusion in the study.
2. Patients who have required treatment with HBIG, or are receiving it at present.
3. Patients from 18 to 70 years of age.
4. The patient agrees to participate and comply with all aspects of the protocol, including the planned blood sample collection, and has signed the informed consent form.

Exclusion Criteria:

1. Presence of HBV DNA or HBeAg indicating virus replication.
2. Patients with known allergies to some component of HB-IVIG, such as sorbitol (e.g. patients presenting intolerance to fructose).
3. Patients with a known background of severe or frequent reactions to products derived from plasma.
4. Patients presenting arterial hypertension that is not clinically controlled.
5. Patients presenting a creatinine value >2 mg/dl, nephrotic syndrome or renal failure.
6. Patients presenting anaemia (haemoglobin < 11 g/dl).
7. Patients being treated with interferon.
8. The patient suffers some acute or chronic medical condition that the investigator believes may interfere with the development or interpretation of the study.
9. The patient is known to abuse of alcohol, opiates, psychotropic agents or other drugs or chemical substances; or has done so in the past 12 months.
10. Pregnant women at the time of inclusion or that may be pregnant in the next 7 months or breast-feeding women.
11. Patients participating in another clinical study, or who have received another investigational product in the last 3 months.
12. Possibility that the patient may be treated with other products containing immunoglobulins in a period of 7 months.
13. Suspicion of conditions that may affect the patient's compliance, including an expected survival of less than 1 year.
14. Any patient that does not have a frozen serum sample previous to the first study medication infusion.
15. Patients with selective IgA deficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-10; Primary Completion 2004-07 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To determine if after 4 months of continuous monthly administration of HB-IVIG Grifols, the anti-hepatitis B antibodies contained in the product reach levels considered as protective, and to assess if these levels are kept constant during 2 more months. | At months 4, 5, and 6

SECONDARY OUTCOMES:
To determine the in vivo recovery of 6 consecutive doses of HB-IVIG Grifols and demonstrate that it remains constant for each dose. | At months 1, 2, 3, 4, 5, and 6
To determine various pharmacokinetic parameters after 6 administrations of HB-IVIG Grifols | At months 1, 2, 3, 4, 5, and 6
To determine the incidence of recurrences during the treatment | At months 1, 2, 3, 4, 5, and 6
To evaluate tolerance to the administration of HB-IVIG Grifols | At months 1, 2, 3, 4, 5, and 6
To confirm the viral safety of the product supervising viral markers | At months 1, 2, 3, 4, 5, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Mas, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Virgen del Rocío, Seville, Sevilla